CLINICAL TRIAL: NCT04161274
Title: Randomized Clinical Trial on Traditional Healing Versus Moist Healing Environment (MHE) Applied to Minor Surgery in the Exeresis of Skin Tags
Brief Title: Randomized Clinical Trial on Skin Tags Approachment.
Acronym: HUM_FIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDIAP JordiGol
Record Dates: First submitted 2019-09-26; First posted 2019-11-13 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2019-07

CONDITIONS: Skin Tags
Keywords: minor surgery procedures; wounds and injuries; moist healing environment; fibroma; nursing; skin diseases
MeSH Terms: conditions — Wounds and Injuries; Fibroma; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traditional method: Electrosurgery (Active Comparator): Local anaesthesia and excision with a scalpel connected to the electric current, according to the voltage. Traditional cure with alcohol/Betadine. Photograph to the lesion before and after the intervention and in each follow-up visit.
  Follow-up visits every 3 days until the lesions cicatrization.
  Interventions: Procedure: Traditional method: Electrosurgery
- Traditional method: Cryotherapy (Active Comparator): Application of liquid nitrogen to cause freezing. Traditional cure with alcohol/Betadine. Photograph to the lesion before and after the intervention and in each follow-up visit.
  Follow-up visits every 3 days until the lesions cicatrization.
  Interventions: Procedure: Traditional method: Cryotherapy
- Traditional method: Silver nitrate (Active Comparator): Excision is made with the scissors and a rod is applied containing silver nitrate with caustic power on the wound.
  Traditional cure with alcohol/Betadine. Photograph to the lesion before and after the intervention and in each follow-up visit.
  Follow-up visits every 3 days until the lesions cicatrization.
  Interventions: Procedure: Traditional method: Silver nitrate
- Moist healing environment (Experimental): Excision is made with the scissors, afterwards pressure, clorhexidine and a hydrocolloid dressing when the skin is dry.
  Photograph to the lesion before and after the intervention and in each follow-up visit.
  Follow-up visits every 3 days until the lesions cicatrization.
  Interventions: Procedure: Moist healing environment method

INTERVENTIONS:
Procedure: Traditional method: Electrosurgery — The patient will be prepared before this technique by removing all metal objects in his possession. The area should be disinfected with a local antiseptic, leaving the area aseptic. Afterwards, perilesional infiltrated local anaesthesia (subcutaneous or intradermal) will be applied. Once the area has been anaesthetised, excision is made with scissors cutting through the most proximal part of the skin tag pendulum and the lesion is coagulated with the handle or knife of the electrocoagulator (previously regulated with the intensity in coagulation mode). The resulting abrasion will form an eschar that will be disinfected with povidone-iodine, and a protective dressing of sterile occlusive gauze bandage will be placed.
  Indications to the patient: the project participant will be instructed to dry the area with povidone-iodine antiseptic and not to expose the area to extreme humidity or sunlight.
  Arms: Traditional method: Electrosurgery
Procedure: Traditional method: Cryotherapy — The patient should be prepared: the area should be disinfected with a local antiseptic, leaving the area aseptic. for a few minutes the tip of an Adson forceps will be introduced in a container with liquid nitrogen until freezing. It will then be applied to the most proximal part of the skin tag pendulum until it is observed that the frostbite has reached the base of the lesion and the surface becomes whitish, with a halo of 1-3 mm. When this happens, it will be excise above the frost part in the pendulum. After application, it is disinfected with povidone- iodine and covered with a protective dressing of sterile occlusive gauze plaster. It will then form an eschar. Indications to the patient: the project participant will be instructed to dry the area with povidone-iodine antiseptic and not to expose the area to extreme humidity or sunlight.
  Arms: Traditional method: Cryotherapy
Procedure: Traditional method: Silver nitrate — The patient should be prepared: the area should be disinfected with a local antiseptic, leaving the area aseptic. Excision will be made with scissors of the skin tag cutting through the most proximal part of the skin tag pendulum, then cauterized with the tip of the silver nitrate rod, trying not to apply in the perilesional zone.
  The resulting abrasion will form an eschar that will be disinfected with povidone-iodine, and a protective dressing of sterile occlusive gauze bandage will be placed.
  Indications to the patient: the project participant will be instructed to dry the area with povidone-iodine antiseptic and not to expose the area to extreme humidity or solar rays.
  Arms: Traditional method: Silver nitrate
Procedure: Moist healing environment method — The patient should be prepared: the area should be disinfected with a local antiseptic, leaving the area aseptic. Excision will be made with scissors of the skin tag by cutting through the most proximal part of the pendulum of the skin tag, later it will be disinfected with chlorhexidine and thin hydrocolloid dressing will be placed. Indications to the patient: the project participant will be told not to touch the dressing until the next control after 3 days with the research team. In case of incidents with the dressing (fall of the dressing), the patient will be given a replacement dressing for this purpose and be able to restore it immediately. It is recommended not to expose the area to the solar rays
  Arms: Moist healing environment

SUMMARY:
Skin tags are a benign dermal disease very frequent in the general population. Their exeresis is indicated in case of discomfort of the affected person (usually because of friction or increase in size). In the minor surgery guidelines, their extraction is recommended with cryotherapy, electrocoagulation or shaving with cauterization of silver nitrate (traditional healing techniques).

This randomized clinical trial proposes its extraction with a non before referenced technique in the manuals of minor surgery and that is nowadays applied with very good outcomes in the domain of pressure ulcers, chronic wounds and, in recent years, in acute wounds; the moist healing environment. Therefore, the investigators propose the surgical exeresis of the fibroid in the most proximal part of the pendulum with the subsequent placement of a thin hydrocolloid dressing.

The objective of this trial is to compare the traditional healing with the moist healing environment in minor surgery, analyzing costs, time invested by the professional, healing time and their respective complications.

Expected results: faster healing and lower cost are expected with the new technique. By contrast, more complications are expected in the techniques of cryotherapy and silver nitrate.

Applicability / Relevance: it is a common pathology usually treated in the minor surgery office or routine visit. Therefore, it can show us which treatment leads to fewer complications for the patient and which is more cost-efficient for the health system.

DETAILED DESCRIPTION:
Study variables:

* Sex: Dichotomous qualitative variable: woman/man. Clinical history collection.
* Age: Discrete quantitative variable in years from the date of birth included in the clinical history.
* Family history. Dichotomous qualitative variable: yes/no. According to the interview with the participant, the family history of first and second degree skin tags will be considered.
* Location of the lesion. Qualitative variable categorized in 6 items: Trunk/ armpit/ neck/ inguinal/ upper extremity/ lower extremity.
* Diabetes Dichotomous qualitative variable: yes/no. According to conditioning factors and problems in the clinical history and interview with the participant. There are studies that relate insulin resistance with the presence or not of skin tags 37, 38. To be able to study if the results obtained are independent of the variable of suffering from DM.
* Cost: Continuous quantitative variable, expressed in euros. The cost will include the performance of the technique in the first minor surgery visit, the post-surgical cures and the follow-up visits. The standardized cost of each of the interventions has been calculated according to the different techniques for approaching skin tag, from the prices published in DOGC 6326 of 1 March 2013 Resolution SLT/353/2013 of 13 February on the review of public price corresponding to the health services provided by the Institut Català de la Salut. Apart from the price for the minor surgery visit of the different approaches, the price of the follow-up visits has been calculated in case of prolonged healing time of the lesion or the appearance of complications (infection or non-viable tissue...).
* Healing time: Discrete quantitative variable expressed in days. It will be considered 'healing' when the lesion has concluded the phases of inflammation and granulation/epithelialization. It will be the moment when it does not require any cure and lacks non-viable tissue (the days in the remodeling phase in which the participant uses skin care such as moisturizing, sun protection... will not be counted). For the monitoring of this variable, in the follow-up visits, the state of scarring will be evaluated and if it is already healed, it will be asked on what day prior to the visit, the lesion did not need any special cure and lacked non-viable tissue.
* Time invested by the professional: Discrete quantitative variable expressed in minutes. The time invested in each visit will be recorded until it is healed.
* Complications:

Infection: Dichotomous qualitative variable: yes/no. Infection is considered when the wound shows inflammation signs of infection.

* Devitalized tissue: Dichotomous qualitative variable: yes/no. The appearance of slough will be observed.
* Technique: Qualitative variable categorized in 4 items:

  * Dry Cure - Electrocoagulation.
  * Dry Cure - Cryotherapy.
  * Dry Cure - Silver Nitrate.
  * Cure in a moist healing environment.

ELIGIBILITY:
Inclusion Criteria:

* Injuries that, by increasing in size or by rubbing with some element of clothing, cause discomfort for the user (pain, bleeding, ...).
* Only small skin tags (≤0,5x0,5cm) will be accepted for study.
* People who voluntarily agree to enter the clinical trial and sign the Informed Consent.

Exclusion Criteria:

* Immunosuppressed patients: people with immunosuppressive treatments, long-lasting corticoids, chemotherapy or radiotherapy, biological treatments and immunosuppressive diseases such as HIV infection, hematological diseases, transplants... (these people have a compromised immune response and are more susceptible to infections and their complications.
* Patients with anticoagulant treatment: oral anticoagulants antagonists of vitamin K (AVK: acenocoumarol, warfarin) or direct oral anticoagulants (DOACs: apixaban, dabigatran, rivaroxaban, edoxaban).
* According to location: those areas of greater risk of infection due to their location (genital areas) or those areas with aesthetic compromise.
* According to size: in order to ensure the homogeneity of the lesions, large lesions (larger than 0,5x0,5cm) will be discarded.
* Allergic to silver (according to medical history or patient reference).
* Lesions of doubtful diagnosis. Skin tag is a benign lesion but any doubt in its diagnostic classification will be an exclusion criterion in its participation. In these cases, it will be treated according to the centre usual minor surgery protocol for study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Healing time | through study completion, an average of 1 year
  Discrete quantitative variable expressed in days. It will be considered 'healing' when the lesion has concluded the phases of inflammation and granulation/epithelialization. It will be the moment when it does not require any cure and lacks non-viable tissue (the days in the remodeling phase in which the participant uses skin care such as moisturizing, sun protection... will not be counted). For the monitoring of this variable, in the follow-up visits, the state of scarring will be evaluated and if it is already healed, it will be asked on what day prior to the visit, the lesion did not need any special cure and lacked non-viable tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Paloma Fürstenheim Milerud, Principal Investigator — ICS; Gemma Amat i Camats, Principal Investigator — ICS
Locations (1):
- Abs Balaguer, Balaguer, Lleida, Spain